CLINICAL TRIAL: NCT00921440
Title: CT Coronary Angiography: Coronary Flow Quantification Supplements Morphological Stenosis Analysis
Brief Title: Computed Tomography Coronary Angiography (CTCA) and Coronary Flow in Stenosis Analysis
Status: Completed | Type: Observational
Sponsor: University of Cologne (Other)
Collaborators: Dept. of Radiology (Unknown)
Responsible Party: Prof. Dr. med. Barbara Krug, University Hospital of Cologne, Dept. Radiology
Other Study IDs: 22462/2 - 2005-070
Record Dates: First submitted 2009-06-15; First posted 2009-06-16 (Estimated); Last update posted 2009-06-16 (Estimated); Status verified 2009-06

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery; stenosis
MeSH Terms: conditions — Coronary Artery Disease; Constriction, Pathologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The investigators' rationale was to evaluate whether a 64-slice CT scanner allows accurate measurement of computed tomographic changes in coronary artery flow profiles and whether CT flow measurements are suitable for classifying the significance and hemodynamic relevance of a stenosis and thereby supplement as a functional parameter for morphological stenosis analysis.

DETAILED DESCRIPTION:
A total of 50 patients prospectively underwent computed tomography coronary angiography (CTCA) in a multidetector CT scanner (Brilliance 64, Philips) ± 1 day before or after invasive coronary angiography (ICA). Immediately thereafter, 2 radiologists reviewed the imaging data to detect any vessel segments with morphology poorly evaluable by CTCA. A locally constant cyclical measurement was acquired in these coronary arteries in breath-hold technique during the passage of a 50ml bolus of contrast media. For analysis, time-density curves of the bolus passage were registered in the coronary artery and the aorta (internal reference), the up-slopes were determined and correlated with each other. The results were compared with the ICA findings.

ELIGIBILITY:
Inclusion Criteria:

* Clinically known or presumed CAD
* Age > 50 years
* Hospitalization for invasive coronary angiography
* Sinus rhythm
* Written informed consent by the patient to participate in the study after comprehensive presentation of the facts

Exclusion Criteria:

* Age <= 50 years
* Contraindications to contrast media administration (medical history of iodine allergy, nephropathy, latent or manifest hyperthyroidism)
* Arrhythmias
* Dyspnea at rest, acute unstable angina pectoris, acute myocardial infarction
* Pregnancy
* Implanted pacemaker
* Unwillingness of patient to consent to the study

Min Age: 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: people with suspected or known coronary artery disease (CAD)
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2007-08; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Krug, Prof. Dr., Principal Investigator — Dept. of Radiology, University Hospital of Cologne